CLINICAL TRIAL: NCT00713908
Title: Voiding Dysfunction in the Postoperative Period Following Placement of the TVT
Status: Terminated | Type: Observational
Why Stopped: The Co-Principal Investigator has moved and is no longer interested in continuing this study at this site.
Sponsor: University of Rochester (Other)
Responsible Party: Michael K. Flynn, MD, University of Rochester
Other Study IDs: 20430
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2009-12

CONDITIONS: Voiding Dysfunction
Keywords: Voiding dysfunction following TVT placement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate how often women have problems passing their urine (voiding) after TVT (Tension Free Vaginal Tape) surgery. This will help us to better understand normal voiding function after surgery as well as to find factors that may help us predict who will have problems after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stress incontinence, diagnosis must be confirmed by cough stress test or multichannel urodynamics
* Undergoing minimally invasive sling procedure - TVT (by transvaginal or surpapubic approach)
* Must be competent to give informed consent

Exclusion Criteria:

* No diagnosis of stress urinary incontinence
* Undergoing minimally invasive sling procedure by route other than TVT
* Undergoing any other pelvic organ prolapse repair procedures
* Pregnancy
* Known voiding dysfunction preoperatively

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Urogynecology clinic
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2007-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Post-void residual volume | Pre-operative and post-operative periods

SECONDARY OUTCOMES:
2-day voiding diary, uroflow, standardized questionnaires | Pre-operatively and post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Michael K. Flynn, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States